CLINICAL TRIAL: NCT07174700
Title: Prevalence of Internet, Gaming, and Porn Addiction and Their Relation With Increased Stress, Anxiety, and Depression Among Medical Students in the MENA Region, a Multinational Cross-sectional Study
Brief Title: Prevalence of Behavioral Addiction and Its Relation With Psychological Disturbance
Status: Active, not recruiting | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Abdelmonam Mamdouh Abdelmonam Mohamed Ahmed Hagag, Dr, Zagazig University
Other Study IDs: ZU-IRB # 1547/29-July-2025
Record Dates: First submitted 2025-08-26; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Internet Addiction; Gaming Disorder; Porn Addiction
MeSH Terms: conditions — Internet Addiction Disorder | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

INTERVENTIONS:
Other: Questionnaire — An online questionnaire will be used to assess the prevalence of internet addiction, gaming addiction, and porn addiction, and their relation with stress, anxiety and depression

SUMMARY:
Internet usage has increased greatly. It is expected to be more than 4 billion by the end of this year. About 80% of them spend most of their internet time on social media, and are expected by 2026 to be about 50% of the total population to use social media at least once a month. The internet is mainly used to connect with friends, relatives, learn new skills, or for entertainment, such as video gaming. However, with this increasing usage, internet addiction can easily increase.

Internet addiction or pathological internet use is defined as uncontrolled, excessive use of it, with uncontrolled time consuming that can cause distress and impairment. The prevalence of internet addiction varied between regions. A study in the seven countries in Europe reported a prevalence of addiction among adolescents to be 1%, and an additional 12.7% at risk of having addiction. In Turkey, a recent cross-sectional study found a prevalence of 18.3%. In the Middle East, the prevalence varied greatly from 0.9% to 33% among adolescents.

Additionally, internet video gaming is another addictive problem that can affect adolescents. A previous meta-analysis showed that gaming addiction prevalence ranged from 0.9% to 19.9%, with males being higher than females. Also, another study showed a prevalence of about 8.4% among Thailand medical students.

On the other hand, overuse of the internet can lead to an increase in problematic pornography use. Another study found a significant association between increased usage of the internet and pornography addiction (P value: <0.001). Additionally, previous studies showed a prevalence of porn addiction ranging from 3.2% to 16.6%. Also, a negative correlation between education level and porn addiction was observed.

All these behavioral addictions increase depression, anxiety, and stress for addicts. Several cross-sectional studies have assessed the positive correlation between either internet, gaming, or porn addiction, and an increase in anxiety and depression. However, to our knowledge, no single study has assessed these three addictive behaviors together with depression, anxiety, and stress in Arab countries.

Rational Medical students, in particular, use the internet frequently. Students use it in training, faculty assignments, research projects, and so on, which can make them depend greatly on the internet. This potentially can increase their addiction to the internet, subsequently increasing their addiction to video gaming and porn addiction. In the Middle East, few studies have tried to assess the prevalence of internet addiction and its association with increased depression, anxiety, and stress among medical students. Despite that, there is a lack of studies on gaming addiction and porn addiction.

The study aimed to assess the prevalence of internet addiction alongside video gaming and porn addiction among medical students and interns in the Middle East (MENA region). Also, the study aimed to assess the relationship of these three addictive behaviors with each other and their relationship with increased stress, anxiety, and depression among this population.

ELIGIBILITY:
Inclusion Criteria:

* Arabic Medical students and interns
* Studying medicine in the Middle East countries
* Have access to online platforms
* Agree to participate in the study

Exclusion Criteria:

* • Students or interns who refused to participate

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Medical students and interns in the Middle East countries are allowed in the study
Sampling Method: Non-Probability Sample
Enrollment: 4600 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
internet addiction | through study completion, an average of 6 months
  We will use the Internet Addiction Scale (IAT). This scale is a 20-question Likert scale, and each question has six answer scales from 0 to 5 (Not applicable, rarely, occasionally, frequently, often, and always). This makes a range of scores from 0 to 100.
  The participants can be classified into normal usage, mild, moderate, and severe levels of addiction if they score (0-30), (31-49), (50-79), and (80-100), respectively.
gaming addiction | through study completion, an average of 6 months
  We will use the Internet Gaming Disorder Scale-Short-Form (IGDS9-SF) This scale consists of a 9-question Likert Scale. Each question has five answers, scored from 1 to 5. Total score ranges from 9 to 45, with a higher score indicating a higher level of gaming disorder.
porn addicton | through study completion, an average of 6 months
  The Problematic Pornography Consumption Scale (PPCS) will be used, which consists of an 18-question Likert Scale. Each question consists of 7 answers, and their scores range from 1-7. A total score ranges from 18-126, with higher levels indicating a higher level of porn addiction. A 76 score will be used as a cut-off value to indicate a high risk of porn addiction.

SECONDARY OUTCOMES:
Anxiety | through study completion, an average of 6 months
  The GAD-7 scale was used to assess the level of anxiety. This scale consists of a 7-question Likert scale, each one has four answers scored from 0-3, making a range of scores from 0-21.
  Students can be classified into minimal, mild, moderate, and severe levels of anxiety if they score (0-4), (5-9), (10-14), and (15-21), respectively.
Depression | through study completion, an average of 6 months
  The PHQ-9 was used to assess the level of depression. A 9-question Likert scale with four answers for each question. Scores range from 0-3, making the range of scores from 0-27.
  Students can be classified into minimal, mild, moderate, moderately severe, and severe levels of depression if they score (0-4), (5-9), (10-14), (15-19), and (20-27), respectively.
Stress | through study completion, an average of 6 months
  The PSS-10 was used to assess the stress level. A 10-question Likert Scale, and each question has 5 answers, which score from 0-4. A total score ranges from 0-40.
  Students can be classified into mild, moderate, and severe levels of stress if they score (0-13), (14-26), and (27-40), respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University Faculty of Medicine and Affiliated Hospital, Zagazig, Egypt

DOCUMENTS (1):
  • Study Protocol (2025-07-29): https://cdn.clinicaltrials.gov/large-docs/00/NCT07174700/Prot_000.pdf